CLINICAL TRIAL: NCT04871490
Title: Improving Detection and Early Action for HPV-positive Oropharynx Cancer
Acronym: IDEA-HPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Eleni M. Rettig, MD, Principal Investigator, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020P003370
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: HPV Positive Oropharyngeal Squamous Cell Carcinoma
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Group (Other): All eligible participants.
  Interventions: Diagnostic Test: Blood test for HPV DNA

INTERVENTIONS:
Diagnostic Test: Blood test for HPV DNA — All participants will have blood tested for HPV DNA.

SUMMARY:
This study aims to determine whether a blood test for HPV DNA can improve diagnosis of HPV-positive oropharynx cancer (HPV-OPC).

DETAILED DESCRIPTION:
The diagnosis of HPV-OPC is often delayed. In this study, individuals with signs or symptoms potentially related to HPV-OPC, such as unexplained throat pain, tonsil or tongue base asymmetry, or a neck mass, will have their blood tested for circulating HPV DNA. A positive test may indicate that their symptoms are caused by HPV-OPC, and their treating physician will be encouraged to complete all the necessary testing to determine whether this is the case.

ELIGIBILITY:
Inclusion Criteria:

* Neck mass present for >2 weeks with no signs/symptoms of infection
* Neck mass present for >2 weeks with signs/symptoms of infection that did not resolve with antibiotic therapy
* Palatine or lingual tonsillar asymmetry on physical exam
* Palatine or lingual tonsillar asymmetry on imaging, including asymmetric FDG uptake in palatine or lingual tonsils on PET-CT scans
* Unexplained throat pain for >2 weeks that did not resolve with antibiotic therapy

Exclusion Criteria:

* Known diagnosis of HPV-OPC

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of circulating HPV DNA | Test results are returned within 1 week.
  Proportion of participants with circulating HPV DNA detected in their blood.

SECONDARY OUTCOMES:
Predictive value of circulating HPV DNA | Long-term follow-up for up to 2 years
  Proportion of participants with positive circulating HPV DNA for whom HPV-OPC is detected
HPV-OPC awareness | At the time of study enrollment
  Awareness of HPV-OPC and other HPV-related malignancies among participants will be assessed by a brief survey
Impact on clinical practice | Within 2-3 weeks of study enrollment
  The proportion of participants for whom clinicla management by the treating clinician is affected by results of the blood test will be measured by a survey sent to treating clinicials

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided